CLINICAL TRIAL: NCT02492464
Title: Double-blind, Randomized Clinical Trial on the Middle-term Effect of the Red Yeast Rice Intake on Endothelial Function and Arterial Stiffness in Subjects With Suboptimal LDL-cholesterol Level in the Context of the Mediterranean Diet
Brief Title: Effects of 10 mg Monacolins on Vascular Health: a Clinical Trial
Acronym: Monasc10_15
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Claudio Borghi, Professor Claudio Borghi, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Monasc10_15
Record Dates: First submitted 2015-06-22; First posted 2015-07-08 (Estimated); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — red yeast rice

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Red yeast rice (Active Comparator): Red yeast rice extract 200 mg, containing 10 mg monacolin K per daily dose, 1 capsule per day, per 6 months
  Interventions: Dietary Supplement: Red yeast rice
- Placebo (Placebo Comparator): Placebo 200 mg (neutral fibre), 1 capsule per day, per 6 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Red yeast rice — 1 capsule to be taken before to sleep, each day, for 6 months
  Arms: Red yeast rice
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
This will be a double-blind randomized clinical trial carried out on subjects with suboptimal control of LDL-cholesterolemia, following a Mediterranean diet, and treated with a red yeast rice extract (containing 10 mg monacolin K per daily dose) or placebo, in order to evaluate the middle-term effects on vascular health evaluated by non invasive methods (Vicorder(R) apparatus)

ELIGIBILITY:
Inclusion Criteria:

* LDL-cholesterol between 130 and 190 mg/dL

Exclusion Criteria:

* Secundary prevention for cardiovascular disease
* Type 2 diabetes
* Assumption of lipid-lowering drug or dietary supplements
* Previous intolerans to read yeast rice including dietary supplements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-05; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Flow mediated dilation (FMD) change from the baseline to the end of treatment period | 6 months

SECONDARY OUTCOMES:
12 hour fasting LDL-cholesterolemia change from the baseline to the end of treatment period | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- S. Orsola-Malpighi University Hospital, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cicero AF, Morbini M, Rosticci M, D''Addato S, Grandi E, Borghi C. Middle-Term Dietary Supplementation with Red Yeast Rice Plus Coenzyme Q10 Improves Lipid Pattern, Endothelial Reactivity and Arterial Stiffness in Moderately Hypercholesterolemic Subjects. Ann Nutr Metab. 2016;68(3):213-9. doi: 10.1159/000445359. Epub 2016 Apr 8. PMID 27055107
- [Derived] Cicero AFG, Fogacci F, Bove M, Veronesi M, Rizzo M, Giovannini M, Borghi C. Short-Term Effects of a Combined Nutraceutical on Lipid Level, Fatty Liver Biomarkers, Hemodynamic Parameters, and Estimated Cardiovascular Disease Risk: A Double-Blind, Placebo-Controlled Randomized Clinical Trial. Adv Ther. 2017 Aug;34(8):1966-1975. doi: 10.1007/s12325-017-0580-1. Epub 2017 Jul 7. PMID 28687937